CLINICAL TRIAL: NCT03217643
Title: Phase 2 Study of Brentuximab Vedotin Associated With CHP Followed by Consolidation With High-dose Therapy / Autologous Stem-cell Transplantation as Frontline Treatment of Patients With Enteropathy-associated T-cell Lymphoma Type 1.
Brief Title: CHP-BV Followed by Consolidation With High-dose Therapy / ASCT as Frontline Treatment of Patients With EATL Type 1.
Acronym: EATL-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imagine Institute (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMIS2015-03
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Enteropathy Associated T-cell Lymphoma
MeSH Terms: conditions — Enteropathy-Associated T-Cell Lymphoma | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brentuximab Vedotin (Experimental): The first part of the treatment (induction) will evaluate BV-CHP. The second part of the treatment (consolidation) will use standard drugs for the treatment of lymphoma. HDT will consist of BEAM conditioning regimen (or BAM if carmustine is not available). Management of HDT/ASCT will be done according to standard practice.
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — The first part of the treatment (induction) will evaluate BV-CHP. The second part of the treatment (consolidation) will use standard drugs for the treatment of lymphoma. HDT will consist of BEAM conditioning regimen (or BAM if carmustine is not available). Management of HDT/ASCT will be done according to standard practice.

SUMMARY:
It has been recently reported that EATL type 1, but not refractory coeliac disease, strongly expressed CD30 and might benefit from brentuximab vedotin. Since the safety profile of the combination brentuximab vedotin and CHP is known and since the role of etoposide as part of induction regimen is not demonstrated, the investigator will assess the efficacy and toxicity of the combination brentuximab vedotin and CHP followed by HDT/ASCT, as frontline treatment of EATL.

DETAILED DESCRIPTION:
Brentuximab vedotin is an anti-CD30 monoclonal antibody conjugated to the cytotoxic drug monomethyl auristatin E. It is currently evaluated in combination with multi-agent chemotherapy as frontline treatment of systemic ALCL (sALCL) and other CD30-positive mature T cell and NK cell lymphomas. Preliminary results of this phase 1 study have been presented at the 2012 ASH Annual Meeting: 26 patients have been treated with combination brentuximab vedotin and CHP. Nineteen of 26 patients had a diagnosis of sALCL and 7 patients had a diagnosis of another mature Tor NK-cell lymphoma (EATL, n=1). The maximum tolerated dose of brentuximab vedotin in combination with CHP was not exceeded at 1.8 mg/kg IV. Adverse events were manageable. All patients achieved an objective response, with 23 patients (88%) achieving a complete response (CR). All 7 non-sALCL patients achieved a CR.

Finally, it has been recently reported that EATL type 1, but not refractory coeliac disease, strongly expressed CD30 and might benefit from brentuximab vedotin. Since the safety profile of the combination brentuximab vedotin and CHP is known and since the role of etoposide as part of induction regimen is not demonstrated, the investigator will assess the efficacy and toxicity of the combination brentuximab vedotin and CHP followed by HDT/ASCT, as frontline treatment of EATL.

ELIGIBILITY:
Main Inclusion Criteria:

1. Histologically confirmed diagnosis of EATL based on criteria established by the World Health Organization (WHO) 2016 Classification of Tumors of Haematopoietic and Lymphoid Tissues.
2. EATL should be CD30-positive with a threshold of 10%.
3. Patients aged ≥ 18 years and < 70 years at the time of study entry.
4. ECOG performance status 0 to 3 at time of study entry.
5. Left Ventricular Ejection Fraction (LVEF) ≥ 45% measured by bidimensional echography or radionuclide ventriculography (MUGA scan).

Main Exclusion Criteria:

1. Participants must not have been treated with any prior chemotherapy for EATL. Patients with previous treatment for refractory celiac disease (i.e., immunosuppressive or immunoregulatory drugs) may be included.
2. Known central nervous system involvement by EATL.
3. Active chronic hepatitis B or C.
4. HIV positive serology.
5. HTLV-1 positive serology.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Evaluate the 2-year progression-free survival | 4 years
  2-year progression-free survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Hermine Olivier, Principal Investigator — Hôpital Necker-Enfants Malades
Locations (1):
- Hopital Necker - Enfants malades, Paris, France

IPD SHARING:
Plan to Share IPD: No